CLINICAL TRIAL: NCT00345618
Title: An International, Multicenter, Randomized, Double-blind, Double-dummy, Parallel Group, Study of 3-month or 6-month Treatment With SSR126517E (3.0 mg s.c. Once-weekly) Versus Oral INR-adjusted Warfarin in the Treatment of Patients With Symptomatic Pulmonary Embolism With or Without Symptomatic Deep Venous Thrombosis
Brief Title: Clinical Study Assessing Idrabiotaparinux Sodium Injections Once-weekly in Pulmonary Embolism Therapeutic Approach
Acronym: CASSIOPEA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EFC6034; EudraCT:2006-001786-42
Record Dates: First submitted 2006-06-27; First posted 2006-06-28 (Estimated); Last update posted 2016-03-21 (Estimated); Status verified 2016-02

CONDITIONS: Embolism; Thrombosis
Keywords: Deep venous thrombosis; pulmonary embolism; anticoagulant drugs
MeSH Terms: conditions — Embolism; Thrombosis; Venous Thrombosis; Pulmonary Embolism | interventions — Warfarin; Avidin; Enoxaparin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Idrabiotaparinux (Experimental): Idrabiotaparinux sodium, 3.0 mg, once-weekly for 3 or 6 months depending on the stratum, after enoxaparin, 1.0 mg/kg, every 12 hours for at least 5 days.
  Avidin, 100 mg, at the discretion of the investigator whenever deemed appropriate and possible (ie, life-threatening bleeding, emergency invasive procedure with the potential of uncontrolled bleeding, or over-dosage).
  Interventions: Drug: Idrabiotaparinux sodium; Drug: Avidin; Drug: Placebo (for warfarin); Drug: Enoxaparin
- Warfarin (Active Comparator): Warfarin, INR-adjusted dose, started 24 hours after the start of enoxaparin, 1.0 mg/kg, every 12 hours for at least 5 days, and continued for 3 or 6 months depending on the stratum.
  Avidin, 100 mg, at the discretion of the investigator whenever deemed appropriate and possible (ie, life-threatening bleeding, emergency invasive procedure with the potential of uncontrolled bleeding, or over-dosage).
  Interventions: Drug: Warfarin; Drug: Placebo (for idrabiotaparinux sodium); Drug: Avidin; Drug: Enoxaparin

INTERVENTIONS:
Drug: Idrabiotaparinux sodium — 0.5 mL pre-filled syringe for 3.0 mg
  Subcutaneous injection
  Other Names: Biotinylated Idraparinux; SSR126517
  Arms: Idrabiotaparinux
Drug: Warfarin — Capsules with 1 or 5 mg for INR-adjusted dose (INR checked at least once a month)
  Oral administration
  Arms: Warfarin
Drug: Placebo (for idrabiotaparinux sodium) — 0.5 mL pre-filled syringe
  Subcutaneous injection
  Arms: Warfarin
Drug: Avidin — 100 mg in 10 mg/mL solution
  Intravenous infusion for 30 minutes
  Other Names: SSR29261
Drug: Placebo (for warfarin) — Warfarin matching capsules
  Oral administration
  Arms: Idrabiotaparinux
Drug: Enoxaparin — Prefilled syringes as locally registered
  Subcutaneous injection

SUMMARY:
Objectives are to evaluate whether idrabiotaparinux sodium (SSR126517E) is as least as effective as a standard warfarin treatment to prevent recurrence of venous thromboembolic events (VTE) in patients with symptomatic pulmonary embolism (PE) with or without symptomatic deep venous thrombosis (DVT) and to assess its safety (bleedings) versus warfarin.

DETAILED DESCRIPTION:
Treatment with a therapeutic dose of any low molecular weight heparin (LMWH) or unfractioned heparin (UFH) or fondaparinux is allowed only within the 36 hours immediately preceding randomization. Randomization is performed as soon as the diagnosis of PE (and DVT if concomitant suspected symptomatic DVT) is confirmed.

Allocation to treatment is done centrally by Interactive Voice Response System (IVRS) and stratified by (1) center, (2) intended treatment duration, ie, 3 months or 6 months. At randomization, the planned duration of treatment (3 or 6 months) is prespecified by the Investigator and determined on the assessment of risk of VTE recurrence. Participants are randomized to either idrabiotaparinux + placebo of warfarin, or warfarin + placebo of idrabiotaparinux, with an initial treatment of at least 5 days with enoxaparin in both treatment groups.

Participants in the 3-month stratum have an additional 13-week observational period after cessation of study treatment. Participants in the 6-month stratum have a 13-week up to 26-week observational period.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic pulmonary embolism with or without symptomatic deep vein thrombosis

Exclusion Criteria:

* End stage renal failure, hepatic failure, uncontrolled hypertension;
* Active bleeding or high risk for bleeding;
* Pregnancy or childbearing potential without proper contraceptive measures, threatened abortion.
* Breastfeeding.
* Known allergy to idraparinux or idrabiotaparinux, avidin or egg proteins;
* hypersensitivity to warfarin, enoxaparin, heparin or pork product; or any other contraindication listed in the labelling of warfarin or enoxaparin;
* Indication of prolonged anticoagulation therapy for other reason than PE;
* Life expectancy < 6 months;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3202 (Actual)
Dates: Start 2006-06; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Recurrence of symptomatic, fatal or not, VTE (PE or DVT) as confirmed by a Central Independent Adjudication Committee (CIAC) | 3 months

SECONDARY OUTCOMES:
Recurrence of symptomatic, fatal or not, VTE (PE or DVT) as confirmed by a Central Independent Adjudication Committee (CIAC) | 6 months
Incidence of any clinically relevant bleeding as classified by the CIAC (ie, major bleeding and other clinically relevant non major bleeding) | 3 months, 6 months and 3- to 6-month post-treatment follow-up

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (38):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Buenos Aires, Argentina
- sanofi-aventis Australia & New Zealand administrative office, Macquarie Park, New South Wales, Australia
- Sanofi-Aventis Administrative Office, Vienna, Austria
- Sanofi-Aventis Administrative Office, Minsk, Belarus
- Sanofi-Aventis Administrative Office, Diegem, Belgium
- Sanofi-Aventis Administrative Office, São Paulo, Brazil
- Sanofi-Aventis Administrative Office, Sofia, Bulgaria
- Sanofi-Aventis Administrative Office, Laval, Canada
- Sanofi-Aventis Administrative Office, Santiago, Chile
- Sanofi-Aventis Administrative Office, Shanghai, China
- Sanofi-Aventis Administrative Office, Bogotá, Colombia
- Sanofi-Aventis Administrative Office, Zagreb, Croatia
- Sanofi-Aventis Administrative Office, Prague, Czechia
- Sanofi-Aventis Administrative Office, Hørsholm, Denmark
- Sanofi-Aventis Administrative Office, Cairo, Egypt
- Sanofi-Aventis Administrative Office, Tallinn, Estonia
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Athens, Greece
- Sanofi-Aventis Administrative Office, Mumbai, India
- Sanofi-Aventis Administrative Office, Netanya, Israel
- Sanofi-Aventis Administrative Office, Milan, Italy
- Sanofi-Aventis Administrative Office, México, Mexico
- Sanofi-Aventis Administrative Office, Gouda, Netherlands
- Sanofi-Aventis Administrative Office, Lysaker, Norway
- Sanofi-Aventis Administrative Office, Lima, Peru
- Sanofi-Aventis Administrative Office, Makati City, Philippines
- Sanofi-Aventis Administrative Office, Warsaw, Poland
- Sanofi-Aventis Administrative Office, Porto Salvo, Portugal
- Sanofi-Aventis Administraive Office, San Juan, Puerto Rico
- Sanofi-Aventis Admnistrative Office, Moscow, Russia
- Sanofi-Aventis Administrative Office, Brastislava, Slovakia
- Sanofi-Aventis Administrative Office, Midrand, South Africa
- Sanofi-Aventis Administrative Office, Barcelona, Spain
- Sanofi-Aventis Administrative Office, Bromma, Sweden
- Sanofi-Aventis Administrative Office, Istanbul, Turkey (Türkiye)
- Sanofi-Aventis Administrative Office, Kiev, Ukraine
- Sanofi-Aventis Administrative Office, Guildford Surrey, United Kingdom

REFERENCES:
- [Result] Buller HR, Gallus AS, Pillion G, Prins MH, Raskob GE; Cassiopea Investigators. Enoxaparin followed by once-weekly idrabiotaparinux versus enoxaparin plus warfarin for patients with acute symptomatic pulmonary embolism: a randomised, double-blind, double-dummy, non-inferiority trial. Lancet. 2012 Jan 14;379(9811):123-9. doi: 10.1016/S0140-6736(11)61505-5. Epub 2011 Nov 28. PMID 22130488